CLINICAL TRIAL: NCT07385729
Title: The Effect of Video-Assisted Instruction on Central Venous Catheter Application Skills, Anxiety, and Satisfaction in Nursing Students: A Randomised Controlled Trial
Brief Title: Effect of Video-Assisted Instruction on Central Venous Catheter Skills in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ATAUNI-CVC-VIDEO-RCT-
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Central Venous Catheter Care; Nursing Education
Keywords: Video-assisted instruction; Central venous catheter care

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either a video-assisted education group or a traditional education group and followed in parallel throughout the study period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation during skill evaluation and data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Assisted Instruction Group (Experimental): Participants received standard theoretical and laboratory-based instruction plus video-assisted training on central venous catheter blood collection, medication administration, and dressing care.
  Interventions: Other: Video-Assisted Instruction
- Traditional Instruction Group (Active Comparator): Participants received standard theoretical and laboratory-based instruction without video-assisted training.
  Interventions: Other: Traditional Education

INTERVENTIONS:
Other: Video-Assisted Instruction — Video-Assisted Instruction Group
  Arms: Video-Assisted Instruction Group
Other: Traditional Education — Traditional Instruction Group
  Arms: Traditional Instruction Group

SUMMARY:
This study aimed to evaluate the effect of video-assisted instruction on central venous catheter (CVC) care skills, anxiety levels, and satisfaction among first-year nursing students. Central venous catheter care requires advanced psychomotor skills and is often associated with anxiety during training.

In this randomized controlled trial, nursing students were assigned to either a video-assisted education group or a traditional education group. Both groups received standard theoretical instruction and laboratory demonstrations. In addition, the intervention group had access to short instructional videos demonstrating blood collection, medication administration, and dressing care related to CVCs.

The primary outcome was students' psychomotor skill performance assessed using an objective structured clinical examination (OSCE). Secondary outcomes included students' state anxiety levels and satisfaction with the training method. The findings of this study are expected to contribute to evidence-based strategies for improving psychomotor skill acquisition in nursing education.

DETAILED DESCRIPTION:
Nursing education aims to equip students with cognitive, affective, and psychomotor competencies necessary for safe and effective clinical practice. Among these competencies, psychomotor skills related to central venous catheter (CVC) care are complex, technically demanding, and frequently associated with increased anxiety among nursing students. Difficulties in skill acquisition may negatively affect students' confidence and clinical performance.

Video-assisted instruction has emerged as an innovative educational method that allows learners to observe clinical procedures repeatedly, supports self-paced learning, and facilitates the transfer of theoretical knowledge into practice. However, evidence regarding the effectiveness of video-assisted instruction on CVC-related skills, anxiety, and satisfaction remains limited.

This study was designed as a randomized controlled trial conducted at the Faculty of Nursing of Atatürk University between May and July 2024. First-year nursing students who met the inclusion criteria were randomly assigned to either an intervention group or a control group. Both groups received standard theoretical education and laboratory-based demonstrations on CVC care as part of the Fundamentals of Nursing course.

In addition to standard education, students in the intervention group were provided with access to short instructional videos demonstrating CVC blood collection, medication administration, and dressing care. These videos were designed to present each procedure step-by-step and were aligned with the skill evaluation criteria used in the study. The control group did not receive video-based instruction during the study period.

The primary outcome of the study was psychomotor skill performance related to CVC care, assessed using an objective structured clinical examination (OSCE) and a validated CVC Care Skill Evaluation Form. Secondary outcomes included students' state anxiety levels measured using the State Anxiety Inventory and satisfaction with the training method assessed using a structured questionnaire.

Data were collected before and after the educational intervention. The study was conducted in accordance with ethical principles, and written informed consent was obtained from all participants. The results of this study are expected to provide evidence on the effectiveness of video-assisted instruction as a supportive educational strategy for improving psychomotor skills in nursing education and informing future curriculum development.

ELIGIBILITY:
Inclusion Criteria:

* First-year nursing students enrolled in the Faculty of Nursing
* Taking the Fundamentals of Nursing course for the first time
* Willingness to participate and providing written informed consent
* Attendance on the days when study data were collected

Exclusion Criteria:

* Students transferred from another program (horizontal or vertical transfer)
* Graduates of health vocational high schools
* Students who withdrew during the study period
* Students absent during data collection or assessment sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Overall CVC Care Skill Performance Score | 1 week after completion of the training
  Overall psychomotor performance in central venous catheter (CVC) care assessed using an Objective Structured Clinical Examination (OSCE).
  Participants receive a single total score ranging from 0 to 100 points, where higher scores indicate better overall performance.

SECONDARY OUTCOMES:
State Anxiety Score (State Anxiety Inventory) | 1 week after completion of the training (immediately before OSCE assessment)
  Total score of the State Anxiety Inventory (range 20-80). Higher scores indicate higher anxiety.
Training Method Satisfaction Score | 1 week after completion of the training (immediately before OSCE assessment)
  Total score of the Satisfaction with Training Methods Questionnaire (range 16-80). Higher scores indicate greater satisfaction.
Blood Collection Skill Score | 1 week after completion of the training (during OSCE assessment)
  Blood collection subscale score of the Central Venous Catheter (CVC) Care Skill Evaluation Form (range 0-36). Higher scores indicate better performance. Assessed during OSCE using the CVC Care Skill Evaluation Form.
Medication Administration Skill Score | 1 week after completion of the training (during OSCE assessment)
  Medication administration subscale score of the CVC Care Skill Evaluation Form (range 0-30). Higher scores indicate better performance. Assessed during OSCE using the CVC Care Skill Evaluation Form.
Dressing Care Skill Score | 1 week after completion of the training (during OSCE assessment)
  Dressing care subscale score of the CVC Care Skill Evaluation Form (range 0-34). Higher scores indicate better performance. Assessed during OSCE using the CVC Care Skill Evaluation Form.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Faculty of Nursing, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No